CLINICAL TRIAL: NCT05932888
Title: A Single Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of QLM3003 in Healthy Adult Chinese Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetic Study of QLM3003 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLM3003-102
Record Dates: First submitted 2023-06-22; First posted 2023-07-06 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLM3003 (Experimental): QLM3003 Single dose
  Interventions: Drug: QLM3003
- QLM3003 Placebo (Placebo Comparator): QLM3003 vehicle Single dose
  Interventions: Drug: QLM3003 Placebo

INTERVENTIONS:
Drug: QLM3003 — 1%（10g∶0.1g）or 1.5%（10g∶0.15g）or 2%（10g∶0.2g）
  Arms: QLM3003
Drug: QLM3003 Placebo — 1%（10g∶0.1g）or 1.5%（10g∶0.15g）or 2%（10g∶0.2g）(matching corresponding study medication)
  Arms: QLM3003 Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of single ascending (SAD) doses of QLM3003 compared to placebo. Also, pharmacokinetics (PK) of qlm3003 will be evaluated.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the safety and tolerability of single ascending (SAD) doses of QLM3003 compared to placebo. Also, pharmacokinetics (PK) of qlm3003 will be evaluated.Eligible subjects will be assigned to a sequential treatment cohort and randomized to each treatment group (active/placebo ). Subject enrollment will continue into the next cohort after review of the dose safety from the previous dose cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subjects between 18-55 years of age (inclusive), male or female
2. The body mass index (BMI equal to body mass/square of body height) of the subjects ranges from 19 to 26 kg/m2 (inclusive), and males of weight not less than or equal to 50 kg, females of weight not less than or equal to 45 kg.
3. Subjects have no sperm donation, egg donation plan, no pregnancy plan and voluntarily take effective contraceptive measures from 14 days before signing the informed consent form to 30 days after the last dose of investigational product;
4. The subjects understand and comply with the study requirements, voluntarily participate in the study and sign the informed consent form.

Exclusion Criteria:

1. Patients who are allergic to the investigational product or its preparation ingredients, or have previous allergic diseases, history of drug allergy, history of skin allergy, or known to be hypersensitive;
2. Patients with clinically relevant skin diseases that are contraindicated in the study or affect the assessment of the administration site at screening, including but not limited to psoriasis, eczema, acne, atopic dermatitis, dysplastic mole, or other skin lesions, and a history of skin cancer;
3. Skin conditions affecting the assessment of the study drug such as ulceration, injury, sunburn, redness and swelling, rash, or abnormal fever, tattoos, birthmarks, skin scars, skin perforations, skin infections on the skin of the target application area at screening and before administration, or disagreeing to removing the hair on the skin of this site;
4. Pregnant or lactating women, and those who cannot use one or more non-drug contraceptive measures during the trial;
5. Patients who have difficulty in collecting blood or cannot tolerate venipuncture, and have a history of fainting needle halo;
6. Those who have special requirements for diet and cannot abide by the unified diet;
7. Excessive consumption of tea, coffee or caffeinated beverages, or consumption of grapefruit, or xanthine-rich foods or beverages within 14 days before screening, or inability to stop consumption of xanthine-rich foods or beverages, or grapefruit or pomelo and products containing grapefruit or pomelo ingredients within 48 hours before dosing and during the trial;
8. Patients who smoked more than 5 cigarettes or the same amount of tobacco daily for 3 months before screening and could not stop using any tobacco products during the trial;
9. Regular drinkers within 6 months before screening, i.e., those who drank more than 14 units of alcohol per week or could not stop using any alcohol-containing products during the trial; or those who took any alcohol-containing products within 48 hours before the first dose, or those who tested positive for alcohol breath before randomization;
10. Drug abusers or those who have used soft drugs within 3 months before screening or hard drugs within 1 year before screening or those who have positive drug abuse screening before randomization;
11. Blood donation or massive blood loss, receiving blood transfusion or using blood products within 3 months before screening;
12. Any surgical procedure within 30 days prior to Screening or planned during the study and within 30 days after the end of the study;
13. Patients who have received any live vaccines within 30 days before screening or need to receive live vaccines during the study;
14. Use of any drug that inhibits or induces hepatic metabolism of the drug within 30 days before screening;
15. Patients who have taken any drug or health product within 14 days before screening;
16. Patients who have participated in and used any drug or medical device clinical trials within 3 months before screening, or within 5 half-lives of other investigational drugs before screening;
17. Patients with previous serious or clinically significant diseases or abnormalities at screening, including but not limited to cardiovascular system, nervous system, respiratory system, blood and lymphatic system, digestive system, immune system, liver, kidney, metabolism and bone system diseases or psychiatric diseases or history of malignant tumors;
18. Abnormal vital signs or clinically significant abnormalities in physical examination, ECG and laboratory tests (subject to the judgment of the clinical study physician);
19. Patients with active tuberculosis suggested by clinical symptoms, signs, laboratory tests or chest radiography at screening;
20. Patients whose white blood cell count, neutrophil count, lymphocyte count or hemoglobin in blood routine examination exceed the normal reference range and have clinical significance judged by the investigator;
21. May increase study-related risks, may interfere with interpretation of study results, or, in the judgment of the investigator, make the investigator and/or sponsor unsuitable for enrollment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-25 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence (severity and causality) of any local and systemic adverse events | 8 days
  adverse events

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of QLM3003 | 8 days
  Cmax
Area Under the Plasma Concentration-Time Curve From 0 to t of QLM3003 | 8 days
  AUC0-t
Area Under the Plasma Concentration-Time Curve From 0 to infinity of QLM3003 | 8 days
  AUC0-∞

CONTACTS AND LOCATIONS:
Overall Officials: guoping Yang, doctor, Study Director — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China